CLINICAL TRIAL: NCT07337057
Title: PROMs in Implant Dentistry: Development of a Dental Implant Standard Set
Brief Title: DEntal implaNt Set: Development and Implementation of a Standardized Outcome Set in Implant Dentistry
Acronym: DENS
Status: Recruiting | Type: Observational
Sponsor: Erasmus Medical Center (Other)
Collaborators: University of Santiago de Compostela (Other); University Medical Center Groningen (Other)
Responsible Party: Principal Investigator, Dr. Justin Pijpe, Principal Investigator, Oral Maxillofacial Surgery Department, Erasmus Medical Center
Other Study IDs: MEC-2023-0688; 1661-2022 (Other Grant/Funding Number: International Team for Implantology (ITI))
Record Dates: First submitted 2025-12-02; First posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Tooth Loss / Rehabilitation
Keywords: Dental implants; Patient reported outcome measures; Core outcome set; Implant dentistry; Peri-implant health
MeSH Terms: conditions — Tooth Loss

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 18 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Implant Group: Patients (18 years and older) that require implants for tooth rehabilitation after loss of tooth/teeth..
  Interventions: Device: Implantology

INTERVENTIONS:
Device: Implantology — Implantology is a branch of dentistry focused on the placement and maintenance of dental implants, which are artificial tooth roots made typically from titanium. These implants are surgically inserted into the jawbone to support crowns, bridges, or dentures, providing a stable and long-lasting solution for missing teeth. Implantology involves careful planning, surgical procedures, and prosthetic restoration, often requiring collaboration between dental specialists. It aims to restore function, aesthetics, and patient quality of life.

SUMMARY:
Rationale Over the past decades, the placement of dental implants and prosthetic rehabilitation has revolutionised dentistry overwhelmingly. It is generally regarded as a safe and reliable method due to the high predictability and survival rates. Survival of suprastructure and implant, health status of the peri-implant tissues and radiographic peri-implant marginal bone loss are commonly used criteria to assess the implant treatment outcome. Although this way of treatment evaluation is important to develop and deliver safe dental implants, it does not provide sufficient information for the development of value-based healthcare.

With this new approach of health outcome measurement, in which patient reported outcomes and clinical outcomes are combined, new definitions of success are created that transform dental implant health care by informed decision making, quality improvement and reducing costs. If dentists and oral surgeons make treatment decisions based on this comprehensive health outcome, patients are more likely to receive high quality care and payers only pay for services that achieve results. Therefore, the development of an implant dentistry specific question set, a Dental Implant Standard Set, capturing both the clinicians' and patients' perspective of implant-related health outcomes is of utmost clinical relevance.

Objective(s) A combination of patient-reported outcomes and clinical health outcomes in a Dental Implant Standard Set enables clinicians to evaluate care delivery and to compare performance in a comprehensive and meaningful way. Therefore, the main aim for this project is to implement a workable Dental Implant Standard Set for the dental implant professional to monitor and improve clinicians and patients' perception of peri-implant health following dental implant treatment, and to monitor and improve the performance of dental implant practice as a whole.

Study type This is a prospectively designed multicenter cohort study including 30 dental practices in the Netherlands and Spain

Study population A total of 1000 consecutive patients will be included by the participating dental practices within 12 months.

Questionnaires regarding the clinical outcomes are administered to the dentists providing the dental implant care. PROMs are administered to the participating patients.

Generally, patients aged 18-70 years that have an indication for implant supported fixed single or multiple tooth replacement or implant-supported removable prosthesis are eligible to participate.

Methods the questionnaires are administered to the participating dentist (for clinical outcomes) and patients (Patient Reported Outcome Measures (PROMs) in combination with the collection of clinical and case mix variables at 6 time points: before and at implant placement, at prosthesis placement and 10-12 months after implant placement. The PROMs is administered via a Questionnaire Manager (QM), that is developed by an external company. Within the QM also case mix and clinical data are registered

Burden and risks No risks are involved throughout the study The concise questionnaires to the patients and participating dentist will be a limited burden to the standard dental implant care.

Recruitment and consent Treating clinicians will recruit participants for this project. Clinicians will provide the patient with a brief overview of the study. Participants will receive a digital questionnaire via a link with an informed consent form and contact details (of the principal investigator) for remaining questions.

Data is not open accessible and patient specific data will be anonymously stored.

DETAILED DESCRIPTION:
Background and Rationale:

Dental implant treatment success has traditionally been evaluated using clinical parameters such as implant survival, marginal bone loss, and tissue health from the clinician perspective. However, the shift toward value-based healthcare requires integration of patient-reported outcome measures (PROMs) to capture treatment value from the patient's perspective.

The recently published Implant Dentistry Core Outcome Set and Measurement (ID-COSM) international consensus established essential domains for implant research but lacks a validated, clinically feasible patient-reported outcome instrument. Existing dental PROMs like The Oral Health Impact Profile with 14 items are too general for implant-specific evaluation, while comprehensive tools like the ICHOM Adult Oral Health Standard Set are too lengthy for routine clinical use.

Study Design:

This prospective multicenter cohort study develops and validates the Dental Implant Set (DENS), a patient-reported outcome measure based on ID-COSM domains and items extracted from validated instruments (The Oral Health Impact Profile with 14 items, the Psychosocial Impact of Dental Aesthetics Questionnaire, the Patient Satisfaction Questionnaire with 18 items, the Dental Satisfaction Questionnaire, and the Quality of My Facial Questionnaire are used). The DENS captures four core domains: pathophysiology, implant/prosthesis lifespan, life impact, and functional outcomes.

Technical Implementation:

Data collection occurs through an integrated online platform using GemTracker and LimeSurvey. Participating clinics receive secure access credentials and standardized protocols. Patient questionnaires are distributed via secure links prior to appointments, with alternative in-clinic completion available. Clinical data entry occurs immediately post-appointment.

Validation Framework:

Psychometric evaluation includes internal consistency reliability (Cronbach's alpha), construct validity through confirmatory factor analysis, convergent validity via correlations with clinical parameters, and known-groups validity comparing patient subgroups. Test-retest reliability assessment occurs between stable timepoints.

Multicenter Design:

Approximately 30 dental implant clinics across Netherlands and Spain participate, each recruiting 50-60 patients. This design ensures diverse patient populations and practice settings while maintaining standardized data collection protocols through investigator calibration meetings.

Follow-up Schedule:

The study follows natural implant treatment phases with assessments at baseline (pre-implantation), 1-2 weeks post-implantation (surgical healing), 3 months post-implantation (tissue maturation), 3 months post-loading (initial functional adaptation), and 10 months post-loading (mature functional outcomes). This timeline aligns with standard implant care protocols.

Quality Assurance:

Standardization is maintained through investigator calibration, protocol training, and real-time data monitoring. Missing data patterns and completion rates are tracked to assess implementation feasibility. The pseudonymized data structure ensures patient privacy while enabling comprehensive analysis.

Expected Outcomes:

The validated DENS will provide a standardized, clinically feasible tool for routine implant outcome assessment, enabling benchmarking between practices, quality improvement initiatives, and value-based healthcare implementation in implant dentistry.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-70 years
* Indication for implant-supported fixed single or multiple tooth replacement
* Indication for implant-supported removable prosthesis
* Immediate implant placement cases
* Implant placement after implant failure

Exclusion Criteria:

* Inadequate oral hygiene
* Physical inability
* Pregnancy
* History of radiotherapy in head and neck region
* Language barriers
* Patients requiring soft tissue grafts prior to dental implant placement
* Patients requiring bone augmentation with harvesting autogenous bone from intraoral sites prior to dental implant placement

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients aged 18-70 years that have an indication for implant supported fixed single or multiple tooth replacement or implant-supported removable prosthesis are eligible to participate in this study. This study will also include patients with immediate implant placement and implant placement after implant failure.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-06-24 (Actual); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Patient-reported outcomes measures | Follow up from baseline (pre-implantation), 1-2 weeks post-implantation (surgical healing), 3 months post-implantation (tissue maturation), 3 months post-loading (initial functional adaptation), and 10 months post-loading
  1. Feasibility of DENS Implementation
  Measure: Completion rate percentage across all timepoints Time Frame: Baseline, 1-2 weeks post-implantation, 3 months post-implantation, 3 months post-loading, 10 months post-loading Description: Percentage of enrolled patients completing DENS questionnaire at each timepoint. Target ≥80% completion rate for clinical implementability.
Internal Consistency Reliability | Follow up from baseline (pre-implantation), 1-2 weeks post-implantation (surgical healing), 3 months post-implantation (tissue maturation), 3 months post-loading (initial functional adaptation), and 10 months post-loading
  Measure: Cronbach's alpha coefficient for DENS domains Time Frame: At study completion (10 months post-loading) Description: Internal consistency reliability based on ID-COSM domains. Target α ≥0.7 for acceptable reliability.

SECONDARY OUTCOMES:
Secondary outcome measures | Follow up from baseline (pre-implantation), 1-2 weeks post-implantation (surgical healing), 3 months post-implantation (tissue maturation), 3 months post-loading (initial functional adaptation), and 10 months post-loading
  DENS Questionnaire Validation: Test-Retest Reliability
  Measure: Intraclass correlation coefficient (ICC) Time Frame: Between baseline and 1-2 weeks post-implantation (clinically stable period) Description: Temporal stability of DENS scores in patients without complications. Target ICC ≥0.7.
Responsiveness to Treatment Phases Measure: Effect sizes (Cohen's d) for DENS domain changes | Time Frame: Follow up from baseline (pre-implantation), 1-2 weeks post-implantation (surgical healing), 3 months post-implantation (tissue maturation), 3 months post-loading (initial functional adaptation), and 10 months post-loading
  Responsiveness to Treatment Phases Measure: Effect sizes (Cohen's d) for DENS domain changes Time Frame: Between treatment phases (implantation, loading, follow-up) Description: Ability of DENS to detect clinically meaningful changes across implant treatment phases.
Convergent Validity Assessment Measure: Correlations between DENS domains and clinical parameters | Time Frame: Follow up from baseline (pre-implantation), 1-2 weeks post-implantation (surgical healing), 3 months post-implantation (tissue maturation), 3 months post-loading (initial functional adaptation), and 10 months post-loading
  Time Frame: 3 months post-implantation, 3 and 10 months post-loading Description: Expected correlations r=0.3-0.7 between DENS life impact scores and clinical measures.

OTHER OUTCOMES:
Pathophysiology Periodontal index | Follow up from baseline (pre-implantation), 1-2 weeks post-implantation (surgical healing), 3 months post-implantation (tissue maturation), 3 months post-loading (initial functional adaptation), and 10 months post-loading
  Pathophysiology: Bleeding on probing, pocket depth, plaque at 3 months post-implant, 3 and 10 months post-loading
Surgical Morbidity | Time Frame: Follow up at baseline (before implant placement), at 1-2 weeks and 3 months post-implant placement.
  Surgical Morbidity: DENS pain/swelling, 5-point Likert (1=Never to 5=Frequently)
Function | Time Frame: Follow up from baseline (pre-implantation), 1-2 weeks post-implantation (surgical healing), 3 months post-implantation (tissue maturation), 3 months post-loading (initial functional adaptation), and 10 months post-loading
  Function: DENS chewing/speech, 5-point Likert (1=Never to 5=Always) all timepoints
Satisfaction Likert Scale | Time Frame: Follow up from baseline (pre-implantation), 1-2 weeks post-implantation (surgical healing), 3 months post-implantation (tissue maturation), 3 months post-loading (initial functional adaptation), and 10 months post-loading
  Satisfaction: DENS treatment satisfaction, 5-point Likert (1=Very Dissatisfied to 5=Very Satisfied) all timepoints
Aesthetics satisfaction | Time Frame: at 3 months and 10 months post-loading of the crown
  Aesthetics: DENS appearance satisfaction, 5-point Likert (1=Very Dissatisfied to 5=Very Satisfied) at 3 and 10 months post-loading
Quality of Life Likert scale | Follow up from baseline (pre-implantation), 1-2 weeks post-implantation (surgical healing), 3 months post-implantation (tissue maturation), 3 months post-loading (initial functional adaptation), and 10 months post-loading
  Quality of Life: DENS life impact, 5-point Likert (1=Never to 5=Always) all timepoints
Comfort Likert Scale | Follow up from baseline (pre-implantation), 1-2 weeks post-implantation (surgical healing), 3 months post-implantation (tissue maturation), 3 months post-loading (initial functional adaptation), and 10 months post-loading
  Comfort: DENS comfort items, 5-point Likert all timepoints
Implant Survival | Time Frame: 1-2 weeks post-implantation (surgical healing), 3 months post-implantation (tissue maturation), 3 months post-loading (initial functional adaptation), and 10 months post-loading
  Implant Survival: Binary complications through 10 months post-loading
Pink Aesthetic score | Time Frame: Follow-up at 3 and 10 months post-loading of the crown
  Pink Aesthetic Score: Professional assessment (0-14) at 3 and 10 months post-loading
Peri-implant Health | Time Frame: 3 months post-implant, 3 and 10 months post-loading of the crown
  Peri-implant Health: Probing depth, bleeding at 3 months post-implant, 3 and 10 months post-loading

CONTACTS AND LOCATIONS:
Overall Officials: Eppo B Wolvius, Prof. PhD. DMD. MD., Principal Investigator — Erasmus Medical Center
Locations (1):
- Erasmus Medical Center, Rotterdam, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided
The IPD sharing plan is currently undecided; the protocol is being submitted to BMJ Open.

REFERENCES:
- [Background] Wittneben JG, Wismeijer D, Bragger U, Joda T, Abou-Ayash S. Patient-reported outcome measures focusing on aesthetics of implant- and tooth-supported fixed dental prostheses: A systematic review and meta-analysis. Clin Oral Implants Res. 2018 Oct;29 Suppl 16:224-240. doi: 10.1111/clr.13295. PMID 30328183
- [Background] van der Meulen MJ, John MT, Naeije M, Lobbezoo F. The Dutch version of the Oral Health Impact Profile (OHIP-NL): Translation, reliability and construct validity. BMC Oral Health. 2008 Apr 11;8:11. doi: 10.1186/1472-6831-8-11. PMID 18405359
- [Background] Torrance GW, Feeny D, Furlong W. Visual analog scales: do they have a role in the measurement of preferences for health states? Med Decis Making. 2001 Jul-Aug;21(4):329-34. doi: 10.1177/0272989X0102100408. PMID 11475389
- [Background] Tan WC, Krishnaswamy G, Ong MM, Lang NP. Patient-reported outcome measures after routine periodontal and implant surgical procedures. J Clin Periodontol. 2014 Jun;41(6):618-24. doi: 10.1111/jcpe.12248. Epub 2014 Apr 21. PMID 24593854
- [Background] Steinmann G, Delnoij D, van de Bovenkamp H, Groote R, Ahaus K. Expert consensus on moving towards a value-based healthcare system in the Netherlands: a Delphi study. BMJ Open. 2021 Apr 12;11(4):e043367. doi: 10.1136/bmjopen-2020-043367. PMID 33846147
- [Background] Slade GD. Derivation and validation of a short-form oral health impact profile. Community Dent Oral Epidemiol. 1997 Aug;25(4):284-90. doi: 10.1111/j.1600-0528.1997.tb00941.x. PMID 9332805
- [Background] Ruiz Henao PA, Caneiro Queija L, Mareque S, Tasende Pereira A, Linares Gonzalez A, Blanco Carrion J. Titanium vs ceramic single dental implants in the anterior maxilla: A 12-month randomized clinical trial. Clin Oral Implants Res. 2021 Aug;32(8):951-961. doi: 10.1111/clr.13788. Epub 2021 Jul 8. PMID 34061402
- [Background] Riordain RN, Glick M, Mashhadani SSAA, Aravamudhan K, Barrow J, Cole D, Crall JJ, Gallagher JE, Gibson J, Hegde S, Kaberry R, Kalenderian E, Karki A, Celeste RK, Listl S, Myers SN, Niederman R, Severin T, Smith MW, Murray Thomson W, Tsakos G, Vujicic M, Watt RG, Whittaker S, Williams DM. Developing a Standard Set of Patient-centred Outcomes for Adult Oral Health - An International, Cross-disciplinary Consensus. Int Dent J. 2021 Feb;71(1):40-52. doi: 10.1111/idj.12604. Epub 2021 Jan 16. PMID 33616051
- [Background] Powell CA, Mealey BL, Deas DE, McDonnell HT, Moritz AJ. Post-surgical infections: prevalence associated with various periodontal surgical procedures. J Periodontol. 2005 Mar;76(3):329-33. doi: 10.1902/jop.2005.76.3.329. PMID 15857064
- [Background] Nielsen HB, Schou S, Bruun NH, Starch-Jensen T. Professional and patient-reported outcomes of two surgical approaches for implant-supported single-crown restoration: 1-year results of a randomized controlled clinical trial. Clin Oral Implants Res. 2022 Feb;33(2):197-208. doi: 10.1111/clr.13883. Epub 2021 Dec 17. PMID 34866250
- [Background] Montero-Martin J, Bravo-Perez M, Albaladejo-Martinez A, Hernandez-Martin LA, Rosel-Gallardo EM. Validation the Oral Health Impact Profile (OHIP-14sp) for adults in Spain. Med Oral Patol Oral Cir Bucal. 2009 Jan 1;14(1):E44-50. PMID 19114956
- [Background] Mareque S, Castelo-Baz P, Lopez-Malla J, Blanco J, Nart J, Valles C. Clinical and esthetic outcomes of immediate implant placement compared to alveolar ridge preservation: a systematic review and meta-analysis. Clin Oral Investig. 2021 Aug;25(8):4735-4748. doi: 10.1007/s00784-021-03986-6. Epub 2021 Jun 7. PMID 34100157
- [Background] Lavrakas, P. J. (2008). Encyclopedia of survey research methods (Vols. 1-0). Thousand Oaks, CA: Sage Publications, Inc.
- [Background] Kunavisarut C, Jarangkul W, Pornprasertsuk-Damrongsri S, Joda T. Patient-reported outcome measures (PROMs) comparing digital and conventional workflows for treatment with posterior single-unit implant restorations: A randomized controlled trial. J Dent. 2022 Feb;117:103875. doi: 10.1016/j.jdent.2021.103875. Epub 2021 Oct 30. PMID 34728252
- [Background] Kragt L, Tiemeier H, Wolvius EB, Ongkosuwito EM. Measuring oral health-related quality of life in orthodontic patients with a short version of the Child Oral Health Impact Profile (COHIP). J Public Health Dent. 2016 Mar;76(2):105-12. doi: 10.1111/jphd.12118. Epub 2015 Sep 2. PMID 26331628
- [Background] Kragt L, Jaddoe V, Wolvius E, Ongkosuwito E. The association of subjective orthodontic treatment need with oral health-related quality of life. Community Dent Oral Epidemiol. 2017 Aug;45(4):365-371. doi: 10.1111/cdoe.12299. Epub 2017 Mar 31. PMID 28370341
- [Background] Jonker BP, Wolvius EB, van der Tas JT, Tahmaseb A, Pijpe J. Esthetics and Patient-Reported Outcomes of Implants Placed with Guided Bone Regeneration and Complete Native Bone: A Prospective Controlled Clinical Trial. Int J Oral Maxillofac Implants. 2020 Mar/Apr;35(2):406-414. doi: 10.11607/jomi.7751. PMID 32142578
- [Background] Jensen C, Raghoebar GM, Kerdijk W, Meijer HJA, Cune MS. Implant-supported mandibular removable partial dentures; patient-based outcome measures in relation to implant position. J Dent. 2016 Dec;55:92-98. doi: 10.1016/j.jdent.2016.10.008. Epub 2016 Oct 18. PMID 27769657
- [Background] Feine J, Abou-Ayash S, Al Mardini M, de Santana RB, Bjelke-Holtermann T, Bornstein MM, Braegger U, Cao O, Cordaro L, Eycken D, Fillion M, Gebran G, Huynh-Ba G, Joda T, Levine R, Mattheos N, Oates TW, Abd-Ul-Salam H, Santosa R, Shahdad S, Storelli S, Sykaras N, Trevino Santos A, Stephanie Webersberger U, Williams MAH, Wilson TG Jr, Wismeijer D, Wittneben JG, Yao CJ, Zubiria JPV. Group 3 ITI Consensus Report: Patient-reported outcome measures associated with implant dentistry. Clin Oral Implants Res. 2018 Oct;29 Suppl 16:270-275. doi: 10.1111/clr.13299. PMID 30328187
- [Background] Tonetti MS, Sanz M, Avila-Ortiz G, Berglundh T, Cairo F, Derks J, Figuero E, Graziani F, Guerra F, Heitz-Mayfield L, Jung RE, Lai H, Needleman I, Papapanou PN, Sailer I, Sanz-Sanchez I, Schwarz F, Shi J, Thoma D. Relevant domains, core outcome sets and measurements for implant dentistry clinical trials: The Implant Dentistry Core Outcome Set and Measurement (ID-COSM) international consensus report. J Clin Periodontol. 2023 May;50 Suppl 25:5-21. doi: 10.1111/jcpe.13808. Epub 2023 May 4. PMID 37143289
- See also: Website for patients and clinicians for information regarding the DENS study — https://www.densresearch.com/